CLINICAL TRIAL: NCT03660137
Title: Magnetic Occult Lesion Localization and Imaging (MOLLI) for Non-palpable Breast Lesions: a Phase 0 Pilot Feasibility Trial
Brief Title: Magnetic Occult Lesion Localization and Imaging (MOLLI)
Acronym: MOLLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Ananth Ravi, Medical Physicist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.1.6
Record Dates: First submitted 2018-03-22; First posted 2018-09-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasms
Keywords: Non-palpable lesion; Localization; Lumpectomy; Breast-Conserving Surgery; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will receive both RSL and MOLLI-guided lumpectomy surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOLLI Localization (Experimental): All patients will be implanted with a MOLLI magnetic seed in addition to the standard-of-care RSL seed. Both systems will be use to localize the respective seeds during the lumpectomy surgery.
  Interventions: Device: MOLLI Localization

INTERVENTIONS:
Device: MOLLI Localization — All patients will also be implanted with an additional MOLLI seed using a specialized introducer needle. A specialized MOLLI probe will be used to find the magnetic seed during the lumpectomy surgery.

SUMMARY:
The proposed trial is a non-randomized, single-arm study examining the technical feasibility and safety of magnetic occult lesion localization and imaging (MOLLI) for Breast Conserving Surgery (BCS), in patients with non-palpable lesions. All patients who have an area of concern in the breast and are identified by their physician as good candidates for BCS are eligible to participate. All patients will undergo standard radioactive seed localization (RSL) for intraoperative surgical guidance concurrently with MOLLI localization. The feasibility trial will take place exclusively at a tertiary care institution (Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada) over a 1-year period. The primary endpoint of this study is to measure the success rate of localizing the MOLLI seed.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION

In contemporary breast cancer management, more than 70% of breast cancer patients are eligible for - and select - breast-conserving therapy (BCS). However, issues with cosmesis, patient experience, and treatment workflow efficiency during the therapeutic process have considerable room for improvement.

BCS consists of a surgical procedure whereby the suspicious tumor and a rim of surrounding normal tissue are removed. Up to one-third of all diagnosed breast cancers are non-palpable,and require some form of pre-operative localization to guide precise surgical excision. Currently, options for localization of non-palpable lesions are suboptimal in terms of patient experience, healthcare system resource utilization, and cost-effectiveness.

One of the most common approaches is radioactive seed localization (RSL). RSL consists of insertion of a small radioactive seed under ultrasound guidance to mark the center and/or borders of the tumor. During the procedure the surgeon uses a hand-held probe to detect the seed and guide surgical excision of the lesion intra-operatively. While RSL is effective the use of a radioactive source is and poses many challenges for patients and staff.

WHAT ARE THE INVESTIGATORS DOING?

The investigative team of surgeons and scientists are examining an alternative approach to BCS called magnetic occult lesion localization and imaging (MOLLI). Analogous to RSL, this procedure involves implantation of a small passive magnetic seed - under ultrasound imaging guidance - directly into or surrounding the tumor; during the procedure the surgeon uses a novel hand-held probe to intra-operatively detect the position of this seed and remove the tumor.

WHY IS THE STUDY BEING CONDUCTED?

MOLLI offers many of the same benefits as RSL but without any radiation. MOLLI also has the potential to be more effective and accurate than other localization methods.

WHAT WILL HAPPEN DURING THE STUDY?

As part of this study, researchers will look at how safe the MOLLI system is in finding the tumor in the participant's breast. The study will also gather information on the participant's experience of having the MOLLI seed placed. Participants will undergo both MOLLI as well as the current standard method, RSL, ensuring that the area of concern will be accurately located and then removed. Approximately 20 women will take part in this study

ARE THERE SIDE EFFECTS?

No side effects are expected from the study treatments. Possible risks associated with using MOLLI include:

* A small risk of bleeding following both visits
* A remote risk of allergic reaction to nickel contained in the MOLLI seeds

WHAT WILL HAPPEN AFTER THE STUDY?

Participants may be contacted by a study team member up to and including 16 weeks (6.5 months) after your procedure to take part in a short telephone questionnaire. The questionnaire should take no more than 5 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older with histologically confirmed unifocal breast cancer and identified as a candidate for BCS, this includes patients with high-risk, premalignant (eg. ductal carcinoma in-situ), or malignant (eg. invasive ductal carcinoma) lesions
* Lesions must be non-palpable and require pre-operative localization for surgical guidance
* Lesions must be between 1-5 cm in maximum dimensions to facilitate placement of seeds (either radioactive or metallic seeds for RSL or MOLLI procedures, respectively), as determined by preoperative breast mammogram and / or ultrasound imaging. Pre-operative MRI is at the discretion of the treating surgeon
* The primary lesion must be visible on ultrasound OR mammogram

Exclusion Criteria:

* Biologically male patients
* Multifocal or multi-centric cancer requiring bracketing or multiple resections for complete excision
* Locally advanced malignant breast cancer
* Any absolute contraindications to BCS
* Pregnancy or lactation
* Unable or unwilling to undergo follow-up at Sunnybrook Health Sciences Centre
* Prior allergy to magnetic seed components (nickel) or any part of the delivery system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
MOLLI Localization Success Rate | Day 3 post marker implantation (during surgical excision)
  The primary goal of this study is to determine the success rate of localizing the MOLLI seed, along with subsequent accurate removal under MOLLI guidance alongside RSL.

SECONDARY OUTCOMES:
Duration of Implantation | Day 0 (during marker implantation)
  The duration of MOLLI marker implantation as carried out by the radiologist.
Specimen Margin Positivity | Day 30
  As reported by anatomical pathology, this metric will evaluate if the excised specimen has negative margins or positive margins.
Re-excision rates at 30 days | Day 30
  Follow-up will determine if patients required a re-excision / re-operation after determination of positive margin status.
European Quality-of-Life Questionnaire - 5 Dimensions (EQ5D) questionnaire to evaluate quality-of-life | Day 0 (baseline), Day 30 (1 month FU)
  EQ5D will evaluate overall quality of life pre- and post-MOLLI surgery. Five questions will be evaluated on a 3 point scale (1 being the worst, 3 being the best). Evaluations will occur prior to implantation and approximately 1 month following surgical excision. The lowest score achievable is 5, the highest score achievable is 15.
Duration of Excision | Day 3 (during surgery)
  The time required to perform surgical excision of the lesion and MOLLI marker.
European Quality-of-Life Visual Analogue Scale (EQVAS) questionnaire to evaluate quality-of-life | Day 0 (baseline), Day 30 (1 month FU)
  EQVAS will evaluate overall quality of life pre- and post-MOLLI surgery. Patients will be asked to rank their overall health on a scale from 0 to 100 (0 being the worst, 100 being the best). The lowest total score is 0, the highest achievable total score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Ananth Ravi, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided